CLINICAL TRIAL: NCT06638437
Title: Prevention of Postsurgical Chronic Pain in Children and Adolescents (PREVENDOL)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Elisabet Sánchez-Rodríguez, Principal Investigator, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PID2020-113869RA-I00; PID2020-113869RA-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Chronic Postsurgical Pain; Chronic Post-surgical Pain; Chronic Postoperative Pain; Chronic Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT group (Experimental): The treatment arm will carry out the CBT preventive program before surgery
  Interventions: Behavioral: Cognitive-behavioral therapy
- Control group (No Intervention): The control arm will not do any preventive program (traditional monitoring)

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — The mobile application will include the following modules:
  1. Psychoeducation: information about what to expect from each phase of the surgical process (i.e., pre-operative, the surgery itself and the post-operative).
  2. Activation control techniques: to teach different activation control techniques such as relaxation, breathing techniques and mindfulness training.
  3. Cognitive restructuring and problem solving: to teach how to change maladaptive pain-related beliefs for more adaptive ones and how to better cope with pain.
  4. Exercises and tasks: to encourage the use of the learning strategies we will offer a number of exercises and tasks
  5. Parent's module: to teach parents about the surgical process and how they can help their children during the process
  Arms: CBT group

SUMMARY:
Chronic postsurgical pain is a health problem with a great societal impact: approximately 20% of all children and adolescents undergoing surgery will develop chronic pain. Importantly, the risk and protective factors that are known (e.g., anxiety, catastrophizing, pain beliefs and pain coping) are modifiable, thus there is a huge potential for the development of both preventive and protective programs to avoid the transition from acute to chronic pain or reduce the impact in the lives of patients when it has already developed.

DETAILED DESCRIPTION:
The main objective of this project is to develop and test a program to prevent the development of chronic postsurgical pain in children and adolescents undergoing surgery in order to improve their quality of life (and that of their families). That program will be implemented in a mobile application.

This proposal will be implemented in 3 phases:

1. Development of the preventive program of chronic postsurgical pain and its implementation in a mobile application
2. Usability test of the mobile application
3. Clinical trial to test the effectiveness of the preventive program

ELIGIBILITY:
Inclusion Criteria:

1. Having to undergo surgery
2. Being between 8 and 18 years old;
3. Having signed the informed consent
4. Having an ASA risk between I and III

Exclusion Criteria:

1. Not being able to understand Spanish
2. Having a physical and/or cognitive impairment that interferes with understanding the instructions and handling of the application (e.g., moderate to severe intellectual disability, blindness)
3. Participating in another clinical trial
4. Undergoing an urgent surgical intervention
5. Being hospitalized in intensive care due to the need for ventilation or hemodynamic support or other complications
6. Having an ASA risk of IV
7. Not having signed the informed consent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (pre and postsurgical) | Baseline (pre); daily for 15 days post-surgery; at 3 and 6 months follow-up
  Pain intensity will be recorded using the 0-10 Numerical Rating Scale, with higher scores indicating greater pain intensity
Pain interference (pre and postsurgical) | Baseline (pre), and at 3 and 6 months after surgery (post)
  Pain intensity will be recorded using the 8-item PROMIS Pediatric Pain Interference Scale, with higher scores indicating greater pain interference. PROMIS measures are scored as T-scores, with a mean of 50 points and an SD of 10.

SECONDARY OUTCOMES:
Change in quality of life | Baseline (pre) and 3 and 6 months follow-up
  Quality of life will be recorded using the Pediatric Quality of Life Inventory (Peds-QL). It has four scales: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Scores range between 0 and 100, with higher scores indicating better quality of life.
Change in functional disability | Baseline (pre) and 3 and 6 months follow-up
  Functional disability will be assessed using the Functional Disability Inventory (FDI). The total FDI score can range from 0 to 60, with higher scores indicating higher levels of disability
Change in anxiety and depressive symptoms | Baseline (pre), before surgery and after the CBT (pre), 3 and 6 months follow-up
  Anxiety and Depressive Symptoms will be recorded using a 4-item PROMIS Pediatric Anxiety Symptoms and a 4-item PROMIS Pediatric Depressive Symptoms, with higher scores indicating greater pain interference. PROMIS measures are scored as T-scores, with a mean of 50 points and an SD of 10.
Change in pain beliefs | Baseline (pre), before surgery and after the CBT (pre), 3 and 6 months follow-up
  Pain beliefs will be assessed using the 35-item Pediatric version of Survey of Pain Attitudes. This questionnaire comprises 7 subscales: Medical cure, Medication, Disability, Emotion, Solicitousness, Control and Exercise. Respondents are asked to report the level of agreement with each item/belief statement on a 3-point Likert scale where 0 means "I do not agree with this", 1 "I am not sure" and 2 "I agree with this". Higher scores in each scale indicate greater confidence in that pain belief.
Change in pain catastrophizing | Baseline (pre), before surgery and after the CBT (pre), 3 and 6 months follow-up
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale for Children (PCS-C). Total scores range from 0 to 52, with higher scores indicating greater pain catastrophizing.
Change in pain coping | Baseline (pre), before surgery and after the CBT (pre), 3 and 6 months follow-up
  Pain coping strategies will be assessed using the 14-item Pain Coping Questionnaire (PCQ). The PCQ has 7 scales: Information Seeking & Problem Solving, Seeking Social Support, Positive Self-Statements, Behavioral Distraction, Cognitive Distraction, Externalizing, and Internalizing/Catastrophizing. Participants are asked to rate how often they use each pain coping response when they are in pain using a 5-point Likert scale (from 1= "Never" to 5 = "Very often") with higher scores indicating greater use of this pain coping strategy.
Change in sleep quality | Baseline (pre); before surgery and after the CBT (pre), daily for 15 days post-surgery; at 3 and 6 months follow-up
  Sleep quality will be assessed using a 0-10 Numerical Rating Scale, with higher scores indicating better sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Sánchez-Rodríguez, Dr., Principal Investigator — University Rovira i Virgili
Locations (3):
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No